CLINICAL TRIAL: NCT01880983
Title: 7202 Mitoferrin-1 Expression in Erythropoietic Protoporphyria (Porphyria Rare Disease Clinical Research Consortium (RDCRC)
Brief Title: Mitoferrin-1 Expression in Erythropoietic Protoporphyria (Porphyria Rare Disease Clinical Research Consortium (RDCRC))
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Porphyria Rare Disease Clinical Research Consortium (Unknown)
Responsible Party: Principal Investigator, Brendan McGuire, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 7202
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Erythropoietic Protoporphyria (EPP)
Keywords: EPP; Bloomer; Porphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Porphyrias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood for lymphoblast transformation

SUMMARY:
The purpose of this study is to identify the biochemical/genetic defects in erythropoietic protoporphyria (EPP). People with EPP have skin sensitivity to sunlight and occasionally develop liver disease. In this study, the investigators hope to learn the nature of the biochemical/genetic defects in EPP because this may help explain the severity of these clinical features.

DETAILED DESCRIPTION:
This study examines the possibility that abnormal expression of the gene mitoferrin-1, which codes for the protein that transports iron in the mitochondria of cells, is a contributing factor to the phenotype in individuals with EPP.

Erythropoietic protoporphyria (EPP) is a human genetic/metabolic disorder in which accumulation of the compound protoporphyrin causes skin sensitivity to sunlight. Some individuals with the disorder also have mild anemia, and a few have hepatobiliary disease. Iron is joined to protoporphyrin to form heme in the mitochondria of cells, under control of the enzyme ferrochelatase. Defects in this process cause the accumulation of protoporphyrin, leading to the biochemical and clinical features of EPP. Abnormalities in the ferrochelatase gene are the major cause of the defect, but do not satisfactorily explain the severity of the phenotype in all subjects. Mitoferrin-1 transports iron to ferrochelatase in the mitochondria of cells for heme formation, and also transports iron for the formation of a compound that keeps ferrochelatase active and stable. Thus, a deficiency of this iron transporter could reduce ferrochelatase activity and contribute to the phenotype in EPP.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in the Longitudinal Study of the Porphyrias with a diagnosis of EPP
2. An individual or parent/guardian who is able to give written informed consent or assent, as appropriate -

Exclusion Criteria:

1. Patient is not enrolled in the Longitudinal Study of the Porphyrias
2. Patient is under the age of 7
3. Patient is cognitively impaired
4. Patient refuses to have blood drawn for establishing lymphoblast line -

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Erythropoietic Protoporphyria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mitoferrin-1 expression | once at study enrollment
  To determine if abnormal mitoferrin-1 (MFRN1) expression contributes to the phenotype of individuals with the genetic/metabolic disorder EPP.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan McGuire, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States